CLINICAL TRIAL: NCT04709822
Title: Remote Delivery of a Brief Visuospatial Interference Intervention to Reduce Intrusive Memories Among Trauma Exposed Women: A Feasibility Study
Brief Title: Remote Delivery of a Brief Visuospatial Interference Intervention to Reduce Intrusive Memories of Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Andri Steinþór Björnsson, Professor, University of Iceland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDVIRMT
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Trauma
Keywords: Intrusive memories
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma exposed women (Experimental): No Intervention: Baseline phase ('A'):
  Measurements collected in a daily diary four times a day (morning, afternoon, evening and night) over one week (number of intrusive memories of trauma). Individual baseline phases will be used as control periods for the primary outcome.
  Experimental: Intervention phase ('B'):
  Measurements collected in a daily diary four times a day during the fifth week after the second intervention session for the primary outcome (number of intrusive memories of trauma).
  Interventions: Behavioral: Visuospatial Interference

INTERVENTIONS:
Behavioral: Visuospatial Interference — Two remote intervention sessions with a researcher including a simple cognitive task (a memory cue and 25 minutes of Tetris game play with mental rotation) alongside accompanying information.
  Participants are instructed that they may continue using the technique self-guided after the first intervention session, and they may opt for additional intervention sessions with remote researcher support (maximum 6 intervention sessions).
  Other Names: Brief cognitive intervention

SUMMARY:
This single case series feasibility study is designed to investigate the feasibility of remote recruitment and delivery of a brief visuospatial interference intervention for decreasing the number of intrusive memories of trauma among trauma-exposed women in Iceland. The current study is an extension on two studies already preregistered (NCT04209283 and NCT04342416) that included some aspects of in-person recruitment and/or intervention delivery (rather than fully remote as we aim for here). The intervention is a simple cognitive task (a memory cue followed by playing the computer game "Tetris") with accompanying information. A within-subjects multiple baseline AB design is used, in that the length of baseline ('A'; no intervention) and intervention ('B') phases vary within-subjects across individual intrusive trauma memories. Participants will aim to complete at least one week of the baseline ('A') phase followed by at least two intervention sessions with a researcher remotely (via telephone or secure video platform). Intervention sessions comprise the simple cognitive task alongside accompanying information presented in the form of brief animated videos (e.g., explaining the target symptom). Participants are instructed that they may continue using the technique self-guided in subsequent weeks, and they may opt for additional intervention sessions with remote researcher support (maximum 6 intervention sessions). Participants will be asked to monitor the occurrence of intrusive memories of trauma in a daily diary. It is predicted that participants will report fewer total intrusive memories in the fifth week after the second intervention session (primary outcome) compared to in the first baseline week. The investigators will also explore whether the frequency of targeted intrusive memories is going to decrease relative to non-targeted intrusive memories. Furthermore, the investigators will explore whether having fewer intrusive memories is related to functioning and/or PTSD, depressive or anxiety symptoms.

DETAILED DESCRIPTION:
Participants complete a total of 3-9 sessions with researchers and sessions will be conducted remotely via telephone or secure video platform (Kara Connect). In the baseline session, questionnaires are administered and the individual intrusive trauma memories will be logged for monitoring their frequency in a daily diary. Participants will record their intrusive memories in the daily diary for at least one week (Week -1) before commencing the intervention. In the first intervention session, a memory will be selected and targeted with the intervention (memory reminder followed by 25 min gameplay with mental rotation). We aim to deliver a second intervention session soon after the first (within approx. one week), targeting the same or a different intrusive memory. Participants are instructed that they may continue using the technique self-guided after the first intervention session, and they may opt for additional intervention sessions with remote researcher support (maximum 6 intervention sessions). Participants continue to monitor the frequency of both targeted and non-targeted intrusive memories in the daily diary throughout Weeks 0-5. Follow-up questionnaires are completed at Week 1, 1-month, and 3-months after the second intervention session. The primary outcome is change in total number of intrusive memories from the baseline week (Week -1) to the fifth week after the second intervention session (Week 5). Participants will also monitor the frequency of their intrusive memories for one week at the 3-month follow-up. The investigators note that the intended time-frames may differ slightly across participants depending on availability and the practicalities of remote delivery.

ELIGIBILITY:
Inclusion Criteria:

* Having experienced at least one criterion A trauma according to the DSM-5
* Having at least two intrusive memories over the previous week
* Reporting being bothered by intrusive memories over the past month (scoring at least a moderate or higher score on PCL-5 item 1)
* Being able and willing to complete 3-9 sessions with researcher
* Being willing to monitor intrusive memories in daily life
* Having access to a smartphone
* Being able to speak Icelandic and read study materials in Icelandic

Exclusion Criteria:

* Current psychotic disorder (determined by the psychotic module on the Mini International Neuropsychiatric Interview (MINI))
* Current manic episode (determined by the bipolar module on the Mini International Neuropsychiatric Interview (MINI))
* Being acutely suicidal (according to the module assessing suicidality on the Mini International Neuropsychiatric Interview (MINI))

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in the total number of intrusive memories of trauma | Week 5 compared to Baseline (Week -1)
  Total number of intrusive memories of traumatic event recorded by participants in a diary daily (morning, afternoon, evening and night) during the fifth week after the second intervention session (Week 5), compared to in the baseline week (Week -1).

SECONDARY OUTCOMES:
Change in the total number of intrusive memories of trauma | Weeks 0-4 and 3-month follow-up compared to Baseline (Week -1)
  Total number of intrusive memories of traumatic event recorded by participants in a diary daily (morning, afternoon, evening and night) during the week of receiving the first two intervention sessions (Week 0), the subsequent four weeks (Weeks 1-4) and a 3-month follow-up, compared to in the baseline week (Week -1).
Unwanted Memories of Trauma (UMT) | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  6 self-rated items measuring the frequency of unwanted memories of the trauma in the previous week on a 7-point scale (from never to many times a day) and the level of distress, nowness, reliving, disconnectedness and whether different triggers are associated with the unwanted memories of the trauma on a 11-point scale (from 0 to 100). High scores indicate more unwanted memories, higher levels of distress/nowness/reliving/disconnectedness and more different triggers.
The Posttraumatic Stress Disorder Checklist 5 (PCL-5) | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  The PCL-5 is a short 20-item self-report scale used to assess the severity of PTSD symptoms corresponding to the DSM-5 criteria for PTSD. Symptoms are rated from 0-4. Higher scores indicate greater severity.
The Patient Health Questionnaire-9 (PHQ-9) | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  The PHQ-9 is a 9-item self-report measure of depression symptoms and the severity of those symptoms. Each item is scored from 0 (i.e., not at all) to 3 (i.e., nearly every day).
The Generalized Anxiety Disorder-7 scale (GAD-7) | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  The GAD-7 is a brief self-report questionnaire designed as a screening tool for symptoms of general anxiety disorder and their severity. Each item is scored from 0 (i.e., not at all) to 3 (i.e., nearly every day).
The Sheehan Disability Scale (SDS) | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  The SDS is a self-report questionnaire which is designed to assess functional impairment across three domains: (1) Work/school, (2) social, and (3) family life. These domains are measured on an 11-point scale which ranges from 0 (i.e., not at all) to 10 (i.e., extremely). The scale will be adjusted to assess impairment associated with intrusive memories.
The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  The WHODAS 2.0 is a 12-item self-rated questionnaire measuring difficulties due to health conditions, including mental or emotional problems (with reference to study event). Scores range from 1 ("none") to 5 ("extremely/cannot do"). The maximum score of the WHODAS is 60; lower scores indicate better functioning.
Impact of intrusive memories on concentration, sleep and stress - ratings | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  Six self-rated items to assess the impact of intrusive memories on concentration, sleep, and stress in the past week. 2 items assessing concentration difficulties in general and due to intrusive memories (11-point scale; high scores indicating more difficulties). 2 items assessing sleep disturbances due to intrusive memories (11-point scale; higher scores indicating more sleep disturbance); and 1 item assessing to what degree intrusive memories affected stress levels (0 = not at all; 10 = affected very much).
Rating of how long intrusive memories disrupted concentration on average | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  One item assessing for how long intrusive memories disrupted concentration on average on a 6-point scale (0 = <1 minute - 6 = > 60 minutes)
Impact of intrusive memories on functioning | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  Two questions assessing the impact intrusive memories have on functioning in daily life. One question is open-ended: "Have the intrusive memories affected your ability to function in your daily life in the past week? If yes, how?" and one question is self-rated: "Have the intrusive memories affected your ability to function in your daily life?" (11-point scale, higher score indicate greater impact on functioning.)
General impact of intrusive memories - ratings | Baseline (Week -1), Weeks 0-5, 3-month follow-up
  Two items both rated on an 11-point scale: 1. "During the last week, how distressing were your intrusive memories (0 = not at all; 10 = very distressing). 2. During the last week, how vivid were your intrusive memories (0 = not at all; 10= very vivid). Administered as part of the intrusive memory diary.

OTHER OUTCOMES:
The Pittsburgh Sleep Quality Index Addendum for PTSD (PSQI-A) | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  A 7 item self-report instrument designed to assess the frequency of disruptive nocturnal behaviors (e.g. acting out dreams, episodes of terror or screaming) common in PTSD. Participants are asked to report symptoms over the past month on a four-point Likert scale, ranging between 0 (never in the past month) and 3 (three or more times each week). The total score ranges from 0 to 21.
Self-rated health rating (SRHR) | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  A single item measuring perceived health status on a seven-point scale (from very good to very bad). Higher scores indicate better health.
Sleep Condition Indicator (SCI-02) | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  Two self-rated items: Item 1 measures the extent of being troubled by poor sleep (with reference to study event) on a 5-point scale (from not at all to very much), and item 2 measures the number of nights in the week with sleep problems on 5 point scale (from 0-1 to 5-7 nights). Each 5-point scale is reverse scored (0 - 4) then summed. Possible total scores range from 0 - 8, with higher values indicative of better sleep.
Sick leave | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  Two bespoke items measuring the total number and the number of full work days of sick leave the participant has taken over the past 4 weeks.
The Time Perspective Questionnaire (TPQ) | Baseline (Week -1), Week 1, 1-month and 3-month follow-ups
  8 self-report items (5-point scale from 1 to 5) measuring time perspective on three subscales: past perspective (items 3, 5, 7), present perspective (items 1, 8) and future perspective (items 2, 4, 6). Item scores for each subscale will be summed. Higher values indicate higher levels of past/present/future time perspective.
The Future Self Questionnaire - shortened version (FSQ) | 3-month follow-up
  A free text response field asking to imagine a future self identity. Then a free text response field to describe a mental image of this identity, 2 items measuring vividness (from 1 "not vivid at all" to 10 "very vivid") and positivity (from 1 "very negative" to 10 "very positive") of that image on a 10-point scale and 1 item measuring the perspective of viewing that mental image ("through own eyes" or "as if seeing oneself") before and after the traumatic event(s). Higher scores on rating scales indicate higher levels of vividness/positivity.
Self-guided intervention adherence - usage of the gameplay intervention in daily life | Week 1, 1-month and 3-month follow-ups
  Two self-report items: "How many times did you manage to play Tetris after you experienced an intrusive memory?" (12-point scale: 0-10 or more than 10). If 1 or more is selected, participant is also asked: "Which of your intrusive memories did you target when you played on your own?" (open-ended question)
Intrusion diary adherence | Baseline (Week -1), Weeks 0-5, 3-month follow-up
  Adherence to the intrusion diary assessed with 1 item: "How accurately did you fill out the diary?" (0= not at all; 10 = very accurately)
Feasibility and acceptability - ratings | 1-month follow-up
  Feasibility and acceptability of the intervention assessed with two self-rated items, "Would you recommend playing Tetris to a friend?" and "Do you consider gameplay to be an acceptable way to reduce the daily frequency of intrusive memories?". Scores could range from 0 - 10 with higher scores indicating greater acceptability/feasibility.
Feasibility and acceptability - open-ended questions | 1-month follow-up
  Feasibility and acceptability of the intervention assessed with two open-ended questions: 1. "How did you feel about playing Tetris after you had an intrusive memory?" 2. "Did you find the intervention helpful? If yes, how?"
Credibility/expectancy scale | Week 0
  Prior to completing the intervention, participants provide 5 ratings of treatment expectancy as well as the degree to which they found the rationale for treatment credible; wording adapted to fit the current study.

CONTACTS AND LOCATIONS:
Overall Officials: Andri Björnsson, PhD, Principal Investigator — University of Iceland
Locations (1):
- University of Iceland, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data is to be made openly available via the Open Science Framework for secondary research.
Time Frame: We aim to make anonymised data openly available after the publication of results in a scientific journal, and for such data to remain available indefinitely.